CLINICAL TRIAL: NCT03005600
Title: Stratification of Risk of Diabetes in Early Pregnancy
Acronym: STRiDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Warwick (Other)
Collaborators: Madras Diabetes Research Foundation (Other); Moi Univeristy (Other)
Responsible Party: Principal Investigator, Dr P Saravanan, Associate Clinical Professor & Honorary Consultant Physician, University of Warwick
Other Study IDs: MRMV0135
Record Dates: First submitted 2016-12-22; First posted 2016-12-29 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Screening, diagnosis, risk stratification, ethnic
MeSH Terms: conditions — Diabetes, Gestational; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Both sites have the capacity for all the necessary measurements. All samples will be temporarily stored in fridge and -20°C freezers after which it will be shifted to -80°C freezers for long term storage.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asian Indian: Recruitment to the Indian cohort will be carried out in urban areas of Chennai and be coordinated from Madras Diabetes Research Foundation (MDRF).
  As a part of their routine care, all pregnant women will undergo regular blood tests at presentation, a dating scan if the last menstrual period is unknown and an ultrasound at 20 weeks of pregnancy for foetal anomalies.
  3400 pregnant women in early pregnancy will be studied in this cohort.
- African: Recruitment to the Kenyan cohort will be based and coordinated from Moi Teaching and Referral hospital (MTRH). The bulk of the recruitment will happen at MTRH with significant contribution from Usain Gisu District hospital (UGDH) and Medi-Heal.
  4000 pregnant women in early pregnancy will be studied in this cohort.

SUMMARY:
Hyperglycaemia in Pregnancy or Gestational Diabetes Mellitus (GDM) is one of the most common obstetric medical conditions which when undetected can cause significant adverse outcomes for the mother and the offspring. Diagnosis is typically made between 24-28 weeks of pregnancy using oral glucose tolerance test (OGTT). Therefore, some damage might have already happened prior to detection. Although universal screening is recommended by many guidelines, this is not uniformly followed across the world, partly because of doubts about cost-effectiveness. Only selective screening is followed based on presence of at least one of the high risk factors (age, BMI, previous history, etc). This strategy can miss up to 50% of GDM. In addition, no data exists in India and Kenya. In low and middle-income countries (LMICs), where majority live in rural settings, the major limitations are difficulty in conducting OGTT, which requires prompt access to laboratory facilities. Combining the clinical and easily analysable biochemical markers (composite risk score) could improve the prediction and if proven, could help to prevent the onset of GDM. Fasting glucose levels (at non-diabetes levels) in early pregnancy could predict future GDM. HbA1c in early pregnancy can be a better marker as it can be done point-of-care and does not require patients to be in a fasting state. The overall objective of the proposed project is to develop a composite risk score to predict GDM in early pregnancy using a combination of easily identifiable risk factors such as age, BMI, family history of Type 2 Diabetes along with HbA1c in Indians and Kenyans. The project will recruit pregnant women in early pregnancy from South India (n=3400) and Western Kenya (n=4000). Contribution of individual risk factors as well as the composite risk score on the risk of developing GDM will be assessed. Detailed health economic analyses will enable policy makers to make informed decision based on local data.

DETAILED DESCRIPTION:
High glucose level in Pregnancy or Gestational Diabetes Mellitus (GDM) is one of the most common medical conditions during pregnancy. When undetected, it can cause significant harm for the pregnant women and her offspring. GDM can affect 5-25% of all pregnant women. It depends on the population and where the boundary is drawn between normal and abnormal glucose levels.

Certain ethnic minority groups are considered at high-risk for developing GDM, including Indians. It is estimated >15% of pregnancies are affected by GDM in India. The immediate risks of untreated GDM are high rates of pre-eclampsia, higher caesarean section rates and psychological effects such as anxiety and depression. Women who develop GDM have a 7-8 times higher life-time risk of type 2 diabetes (T2D). Similarly, the immediate risks to the children are being too big or too small, shoulder damage during labour, low glucose levels or jaundice at birth, difficulty in breathing and in rare cases stillbirth. In the long term, the risk of obesity and T2D is also higher.

The diagnosis of GDM is usually made between 24-28 weeks of pregnancy using a glucose drink test called oral glucose tolerance test (OGTT). Although treatment can improve the outcomes, some of the damage may have already been done before the detection of GDM. Therefore, screening to detect high glucose level in pregnancy seems beneficial. However, there can be harms as well as benefits in screening programmes. Therefore a balance should be achieved between identifying women whose blood glucose level is high enough to cause harm and those with glucose level that would not cause harm. Currently, it is recommended that all pregnant women should be screened for GDM if they belong to a high-risk ethnic population. However, conducting OGTT in India is challenging, as this test requires pregnant women present themselves to a laboratory facility in a fasting state.

In many countries, women are selected for OGTT based on the presence of at least one of the high risk factors such as higher body weight, older age and family history of T2D. However, this selection method can miss up to 50% of women who may develop GDM. The aim of the study is to develop a risk score in early pregnancy based on a combination of these risk factors that can be collected easily along with a simple finger prick average blood glucose test (called HbA1c). The efficiency of different levels of this combined risk score will be tested against the risk of developing GDM in the later part of pregnancy.

Cost effectiveness analysis will also be conducted to identify at what risk level screening can be recommended in India. An accurate score that can safely exclude women at low risk of developing GDM will have significant benefits to the pregnant women. They can be safely reassured. Avoiding the need for OGTT will have significant time and cost benefits. In contrast, if the score identifies them as at high-risk, healthy eating and appropriate life style advice can reduce their risk of developing GDM in later pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women between the age of 18 and 50 years of age

Exclusion Criteria:

* Women presenting beyond 16 weeks of gestation Known Type 1 or Type 2 diabetes
* Severe anaemia defined as haemoglobin (Hb) <8g/L and
* Sickle cell traits, sickle cell anaemia and other genetic Hb variants
* Women on Metformin therapy for anovulation and/or infertility

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The project will be set in and around Chennai (Tamil Nadu, South India) and Eldoret (Western Kenya). Two independent cohorts will be formed, comprising of 3400 and 4000 pregnant women in early pregnancy in India and Kenya, respectively.
Sampling Method: Probability Sample
Enrollment: 7400 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-07 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Development and validation of composite risk score for GDM with the risk factors of interest and/or point-of-care HbA1c | 3 YEARS

SECONDARY OUTCOMES:
Identification and the impact of other novel risk factors on the diagnosis of GDM and other adverse maternal outcomes | 3 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: Ponnusamy Saravanan, FRCP PhD, Principal Investigator — University of Warwick
Locations (2):
- Madras Diabetes Research Foundation, Chennai, Tamil Nadu, India
- Moi University School of Medicine & Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Metadata will be archived following the publication of the study findings as per MRC UK's guidelines